CLINICAL TRIAL: NCT01476462
Title: Second Malignant Neoplasms After Childhood ALL Therapy; An International Ponte di Legno Study
Brief Title: Second Malignant Neoplasms After Childhood ALL Therapy
Acronym: PdL-SMN1
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Nordic Society for Pediatric Hematology and Oncology (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); Dana-Farber Cancer Institute (Other); ALL-BFM Study Group (Network); Dutch Childhood Oncology Group (Other); St. Jude Children's Research Hospital (Other); United Kingdom Children's Cancer Study Group (Other)
Responsible Party: Principal Investigator, Kjeld Schmiegelow, Professor, Rigshospitalet, Denmark
Other Study IDs: PdL SMN Study 1
Record Dates: First submitted 2011-07-13; First posted 2011-11-22 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia; Ponte-di-Legno consortium; Second cancer; Survival
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALL diagnosed 1980-2007: Cases of childhood acute lymphoblastic leukemia (ALL) diagnosed between 1980 and 2007 and included in the clinical trials of the participating ALL study groups

SUMMARY:
Development of a second neoplasm (SMN) during or after therapy for childhood acute lymphoblastic leukemia (ALL) is a rare event generally associated with a poor prognosis. In this international study we analyze subtypes of SMN in relation to their initial leukemia characteristics and treatment, and their subsequent overall survival.

DETAILED DESCRIPTION:
To explore epidemiology, potential risk factors and survival rates of second cancers occurring as the first event in childhood acute lymphoblastic leukemia the involved study groups will collect anonymous data on all such cases diagnosed within the last decades to form a common database with predefined variables comprising the clinical, biological, and cytogenetic characteristics (myeloid neoplasias only) as well as outcome. Furthermore, we will register the clinical, biological, and cytogenetic characteristics of the acute lymphoblastic leukemia as well as type of treatment given.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with childhood acute lymphoblastic leukemia
* Diagnosis of second cancer before December 31st 2007

Exclusion Criteria:

* Uncertainty if the second cancer has emerged from the same original leukemic clone

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study cohort includes all registered cases of second cancers occurring as the first event among children diagnosed with acute lymphoblastic leukemia and treated according to protocol by one of the collaborative groups participating in the present study
Sampling Method: Non-Probability Sample
Enrollment: 642 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pattern of SMN subtypes | At 20 years from diagnosis
  Pattern of the main groups of SMN and their clinical charactiristics
Overall survival by subtype | At 10 years from diagnosis of SMN
  Overall survival by the main SMN subtypes (myeloid malignancies, brain tumors, lymphomas, sarcomas, carcinomas, others)
Risk factors for development of SMN | At 20 years from ALL diagnosis
  Identification of risk factors linked to the interval to SMN, the subtype of SMN, and the survival after. These risk factors are clinical characteristics of ALL or the anti-ALL therapy administered

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D., Principal Investigator — Rigshospitalet, Denmark; Maria G Valsecchi, M.Sci,, Principal Investigator — Dipartimento di medicina clinica e prevenzione, University of Milan, Italy
Locations (1):
- Kjeld Schmiegelow, Copenhagen, Denmark